CLINICAL TRIAL: NCT00763581
Title: Personal Adherence Evaluation of Individuals Receiving Treatment for Bipolar Disorder (PAE in BD)
Brief Title: Personal Adherence Evaluation of Medication Use for Adult Bipolar Disorder Patients
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Martha Sajatovic, MD, Professor of Psychiatry, Case Western Reserve University
Other Study IDs: R34MH078967-01 (NIH); R34MH078967-01 (NIH); R34MH078967 (NIH); DAHBR 96-BHA
Record Dates: First submitted 2008-09-19; First posted 2008-10-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Bipolar Disorder
Keywords: Patient Non-Adherence; Patient Non-Compliance; Patient Nonadherence; Patient Noncompliance; Patient Refusal of Treatment; Treatment Refusal; Refusal of Treatment
MeSH Terms: conditions — Bipolar Disorder; Patient Compliance; Treatment Refusal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will attempt to increase understanding of why bipolar disorder patients do or do not take their medications by conducting in-depth interviews with them.

DETAILED DESCRIPTION:
Disruptive manic and depressive episodes prevent bipolar disorder (BPD) sufferers from living healthy, functional lives. Relapse rates for BPD are high, between 70% and 90%, with approximately half of those relapses occurring in the first 2 years after remission. High rates of relapse and no substantial improvements in illness outcomes for many patients despite advances in drug treatment may be related to a common problem: medication nonadherence. Nine in 10 individuals with BPD have seriously considered medication withdrawal, and one third of individuals with BDP do not take 30% or more of their prescribed medications. The researchers in this study will identify BPD patients who do not take their medications as prescribed and conduct interviews with them. By obtaining an understanding of subjective reasons for medication nonadherence, this study will pave the way for better interventions to ensure BDP patients take the medications that will help them.

Participation in this study will consist of a single visit, lasting between 1.5 and 3 hours. All participants will have a history of medication nonadherence. Participants will be asked to fill out questionnaires and undergo a structured interview with a researcher. The interview will be audio recorded. The questionnaires and interview will assess BPD symptoms, attitudes toward medications, and to what extent patients are taking their medications. Researchers will also measure the number of pills used in participants' prescriptions by counting how many pills are left in each prescription bottle.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of bipolar disorder (BPD) Type I or Type II, as determined by a standardized diagnostic interview, the Mini-International Neuropsychiatric Interview (MINI)
* Demonstrated history of poor medication adherence, as determined by self-report or clinician report. In this study, self-reported treatment nonadherence will be identified with the Tablet Routines Questionnaire (TRQ). Poorly adherent individuals will be defined as those who miss 30% or more of medication within either the past week or past month (those missing 30% or more within past week will be considered to be non-adherent over the past month). Clinician-assessed nonadherence will be identified via a clinician version of the TRQ to identify nonadherence of 30% or more over the past 30 days.
* BPD of at least 2 years' duration
* Treatment with medication to stabilize mood for at least 6 months
* A Clinical Global Impression (CGI-BP) overall bipolar illness score of 4 or higher

Exclusion Criteria:

* Unable or unwilling to participate in psychiatric interviews, as based on the clinical opinion of the investigator or the treating clinician
* High risk of suicide, as seen in factors such as active suicidal ideation, recent suicide attempt, or current suicidal intent or plan
* Inability to speak English
* Receiving treatment involuntarily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty adults (10 men and 10 women) receiving standard outpatient mental health treatment at Connections, a community mental health clinic (CMHC).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Subjective Experience of Medication Interview (SEMI) TAD BD, a qualitative instrument modified from the original SEMI | An average of 4 hours

SECONDARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | An average of 4 hours
Young Mania Rating Scale (YMRS) | An average of 4 hours
Brief Psychiatric Rating Scale (BPRS) | An average of 4 hours
Clinical Global Impression for Bipolar Disorder (CGI-BP) | An average of 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Martha Sajatovic, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- Connections, Cleveland, Ohio, United States